CLINICAL TRIAL: NCT02058082
Title: Randomized Control Trial on the Use of Testicular Versus Ejaculated Spermatozoa for IVF/ICSI on Pregnancy Outcomes for Men With High Sperm DNA Damage
Brief Title: Testicular Versus Ejaculated Spermatozoa for IVF/ICSI in Men With High Sperm DNA Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Kirk Lo, Associate Professor, Division Urology Mount Sinai Hospital, University Toronto, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sperm DNA damage study
Record Dates: First submitted 2014-01-27; First posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Infertility, Male; DNA Damage
Keywords: Failure to Conceive Due to Infertility of Male Partner; DNA Damage
MeSH Terms: conditions — Infertility, Male | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ejaculated sperm (Active Comparator): Intracytoplasmic sperm injection (ICSI) cycles using ejaculated sperm
  Interventions: Procedure: Intracytoplasmic sperm injection
- testicular extracted sperm (Active Comparator): Intracytoplasmic sperm injection (ICSI) cycles using testicular extracted sperm
  Interventions: Procedure: Intracytoplasmic sperm injection

INTERVENTIONS:
Procedure: Intracytoplasmic sperm injection

SUMMARY:
The purpose of this study is to determine whether couples undergoing IVF/ICSI with male factor infertility, specifically with elevated sperm DNA damage, should testicular sperm extraction be utilized to improve their reproductive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* be considered infertile (>1 year of unsuccessful attempts of conception
* Any race
* Male partner with persistent sperm DNA damage, DFI>=30%
* candidates for intracytoplasmic sperm injection (ICSI)

Exclusion Criteria:

* significant female factor infertility contributing to the couple's infertility
* female partner older than 38 years
* male or female patients with genetic abnormalities
* patients unable or unwilling to give consent after properly informed
* couples unsuitable for IVF/ICSI
* male patients in whom testicular procedures were contraindicated

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-06; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Live birth rates | Up to 1 year

SECONDARY OUTCOMES:
sperm DNA damage | Mesaured at baseline, 3 months and on the day of Intracytoplasmic sperm injection (ICSI) procedure
oocyte fertilization rates | at approximately 18 hrs post Intracytoplasmic sperm injection (ICSI)
embryo cleavage rate | Day 3 post oocytes retrieval
blastocyst rate | Day 5 post oocytes retrieval
pregnancy rate | 6 to 8 week ultrasound
  Clinical pregnancy was defined as the ultrasonographic visualization of one or more gestational sacs and fetal heart at the 6 to 8 week ultrasound
rate of spontaneous abortion | after a clinical pregnancy has been established, up to 10 months after procedure
birth defects | 1-year following delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kirk C. Lo, MD, Principal Investigator — MOUNT SINAI HOSPITAL